CLINICAL TRIAL: NCT07220525
Title: Disrupted Sleep and Concurrent Ectopy or Atrial Fibrillation
Acronym: DISCRETE AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 25-43785
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea; Premature Ventricular Contraction (PVC); Atrial Fibrillation (AF); Premature Atrial Contraction
Keywords: Sleep Apnea; Hypoglossal Nerve Stimulation Device; Atrial Fibrillation; Upper Airway Stimulation; Premature Atrial Contraction; Premature Ventricular Contraction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Ventricular Premature Complexes; Atrial Fibrillation; Atrial Premature Complexes; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HGNS 'Off' Case-Crossover Arm (Experimental): On a given day of the 14-day study period, participants may be randomly assigned to turn off/not use their HGNS device during that night of sleep. Participants will not receive the same randomization assignment more than two consecutive days in a row.
  Interventions: Device: HGNS Use Randomized Instructions
- HGNS 'On' Case-Crossover Arm (Experimental): On a given day of the 14-day study period, participants may be randomly assigned to turn on/use their HGNS device during that night of sleep. Participants will not receive the same randomization assignment more than two consecutive days in a row.
  Interventions: Device: HGNS Use Randomized Instructions

INTERVENTIONS:
Device: HGNS Use Randomized Instructions — In this intervention assignment, participants will be instructed to turn off/not use their HGNS device during that night of sleep. HGNS 'on': In this intervention assignment, participants will be instructed to turn on/use their HGNS device during that night of sleep.

SUMMARY:
Whereas the available evidence mostly supports chronic sleep disruption as a risk factor for incident AF, less is known about the near-term risk of a discrete atrial fibrillation (AF) episode following a night of disrupted or poor-quality sleep. This prospective, randomized, case-crossover study aims to examine the acute effects of sleep disruption on clinically relevant cardiac ectopy pertinent to AF.

DETAILED DESCRIPTION:
One hundred patients aged 21 years or older who have a hypoglossal nerve stimulation (HGNS) device implanted for obstructive sleep apnea, without a history of permanent AF, not on Class 1 or 3 antiarrhythmic medications and willing to participate in the study, will be randomized to "off-on" versus "on-off" periods (where "off" is turning off the HGNS device for one night and "on" is turning on the HGNS device), assuring no more than two consecutive days of either device use or not, over the ensuing 14 days. Participants will be fitted with an automatically recording electrocardiographic monitor. The primary endpoint will be the daily number of cardiac ectopic beats, and secondary endpoints: daily number of PACs, daily number of PVCs, and daily presence versus absence of AF episodes ≥ 30 seconds. Primary analyses will employ intention-to-treat principles, examining randomization assignment as the primary predictor.

ELIGIBILITY:
Inclusion Criteria:

* Are age 21 years or older
* Have a HGNS device implanted for obstructive sleep apnea and followed up at UCSF Health
* Are willing to abstain from using the upper airway stimulation device for no more than two consecutive days as instructed over the 14-day trial period
* Able and willing to provide written informed consent

Exclusion Criteria:

* Currently pregnant or trying to get pregnant
* Are currently taking class 1 or 3 anti-arrhythmic medications
* Have a history of permanent AF or expected to have continuous AF throughout the study period
* Have congenital heart disease
* Ventricular pacing >40%
* Are unable to read or sign to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Ectopic beats | 24-hour time period
  Daily number of ectopic beats as recorded with the adhesive heart monitor

SECONDARY OUTCOMES:
Premature Atrial Contractions (PACs) | 24-hour time period
  Daily number of PACs as recorded with the adhesive heart monitor
Premature Ventricular Contractions (PVCs) | 24-hour time period
  Daily number of PVCs as recorded with the adhesive heart monitor
Atrial Fibrillation (AF) | 24-hour time period
  Daily presence of AF ≥30 seconds as recorded with the adhesive heart monitor

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Parnassus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT07220525/Prot_000.pdf